CLINICAL TRIAL: NCT06930924
Title: Evaluation of a Self-help Psychological Intervention to Support Gluten-free Diet Management, Psychological Wellbeing and Quality-of-life in Children and Young People (Aged 7-11) With Coeliac Disease
Brief Title: Supporting Children and Young People to Live Well With Coeliac Disease: A RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: Coeliac UK (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPON-2024-28
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Coeliac Disease; Celiac Disease in Children
Keywords: Coeliac disease; celiac disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parent self-help psychological resource (Experimental): A self-help psychological resource will be provided for parents to use with their CYP in the home. Parents can also attend an online peer support information workshop.
  Interventions: Behavioral: Parent self-help psychological resource
- Wait list control (No Intervention): Parents randomised to the control arm will be put on the waiting list (wait-list controls) to receive the group intervention after they have completed their final follow-up at 5 months.

INTERVENTIONS:
Behavioral: Parent self-help psychological resource — A self-help psychological resource designed alongside families and clinicians, to be delivered to parents of CYP with coeliac disease. The resource will focus on providing psychoeducation on the gluten-free diet, concerns around dietary management, using family's strengths to support dietary management, managing outside the home, and transition to independent management of the gluten-free diet. Parents will also attend a 60-minute online peer support and information workshop
  Arms: Parent self-help psychological resource

SUMMARY:
Managing a strict gluten-free diet is crucial for children and young people with coeliac disease. However, this can have adverse effects on psychological well-being and quality of life. Despite appeals from families, clinicians, and researchers, psychological support is not routinely provided to these families. A feasibility project (NCT06007898) adapted existing self-help psychological resources used for food allergy, gastrointestinal disease, and type one diabetes to cater to families dealing with coeliac disease. This feasibility randomised controlled trial was conducted with 100 families and highlighted the viability and acceptability of this self-help resource. This pilot study was conducted in consultation with caregiver(s), clinicians, and CYP living with coeliac disease. These consultations confirmed a lack of support in this area and the enthusiasm for self-help psychological interventions. We will now run a full randomised controlled trial to evaluate the effectiveness of the intervention for caregiver(s) of CYP with coeliac disease in supporting the appropriate management of the gluten-free diet, alongside psychological wellbeing.

For this trial, 172 families will complete well-being and quality of life questionnaires, along with assessments of their child's gluten-free dietary management. Families will be divided into groups receiving the psychological resources either immediately or after a five-month delay. Follow-up questionnaires will be administered at one, two, and five months for all families, regardless of intervention access. Feedback on the resources and research participation will be gathered. The expectation is that these self-help psychological resources for parents will enhance gluten-free diet management, quality of life for coeliac children and young people, and well-being for parents.

DETAILED DESCRIPTION:
Coeliac disease is a common autoimmune condition in children, estimated to affect 1 in 100 in the UK. Coeliac disease can occur at any age and is treated with a lifelong gluten-free diet. When someone with coeliac disease eats gluten (a protein found in wheat, barley and rye), their immune system attacks itself and causes damage to the gut. If left undiagnosed and untreated long term, the disease can cause complications like growth problems, delayed puberty, tooth enamel defects, iron deficiency anaemia, chronic fatigue and, over time, osteoporosis. The good news is, these potential complications can be avoided with early diagnosis and treatment.

While strict management of the gluten-free diet has been linked to improvements in intestinal damage and quality of life, the relentless behavioural and social demands of detecting gluten is challenging. Often, families report concerns around attending family gatherings, school trips, and eating out at restaurants due to the potential for accidental gluten consumption. To manage these concerns, some families avoid social events entirely, which can affect school attendance and participation in normal childhood activities such as birthday parties and sleepovers. Children and young people (CYP) with coeliac disease have described feeling like a "nuisance" and may experience social stigma associated with their need to eat different food, frustration and isolation, and a higher probability of developing mental health conditions, such as depression, anxiety, or eating disorders.

A large body of research suggests that exposure to parental anxiety increases the risk of similar problems in CYP. CYP can learn that certain situations lead their parents to feel anxious, which may lead to them feeling threatened, and cope (usually by avoidance) in a similar manner. The same appears true for families with coeliac disease, where caregiver(s) with high levels of anxiety, have CYP with higher levels of anxiety. Whilst the gluten-free diet is essential for the management of coeliac disease, it is not enough to only address foods that must that be avoided in coeliac disease. Support must also address how to navigate a gluten-free diet that does not require social isolation and over-restriction. For CYP with coeliac disease, management of the gluten-free diet often relies on the caregiver(s), and so, intervention components must support the whole family system.

Our research team have already developed self-help psychological interventions (interactive websites and books) for families of CYP with food allergy and type one diabetes. We have demonstrated the impact of embedding these interventions alongside routine care for CYP with food allergy, and we are currently testing this approach in type one diabetes. Our findings suggest that these interventions reduce anxiety and increase wellbeing in caregiver(s), as well as their CYP.

We have also completed a pilot RCT of a self-help psychological intervention for families of CYP with coeliac disease (publication in preparation). This pilot study was conducted in consultation with caregiver(s), clinicians, and CYP living with coeliac disease. These consultations confirmed a lack of support in this area and the enthusiasm for self-help psychological interventions. This enthusiasm was reflected in the high participant demand and intervention engagement observed during the pilot study, along with qualitative feedback from families and the NHS Long Term Plan, indicates that self-help psychological interventions for CD are warranted. We will now run a full randomised controlled trial to evaluate the effectiveness of our intervention for caregiver(s) of CYP with coeliac disease in supporting the appropriate management of the gluten-free diet, alongside psychological wellbeing.

ELIGIBILITY:
Inclusion Criteria:

Caregiver(s) with a CYP between 7-11 years of age who report a diagnosis of coeliac disease Willingness to take part in a self-help psychological intervention Participant must have the ability to provide informed consent/assent. Caregiver(s) who consent to the study will still be able to take part, even if their CYP does not provide assent to complete outcome measures

Exclusion Criteria:

Families participating in another intervention-based research will not be eligible Participant identified by clinical team as not appropriate (e.g. undergoing treatment for other complex difficulties) English proficiency unsuitable for participation in self-help psychological intervention and/ or online survey.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The Pediatric Quality of Life scale (parent-report) | Baseline, 1-month, 2-months, 5-months
  Parent reported measure to assess children's quality of life. Scores are converted to a 0 to 100 scale, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Knowledge about the gluten-free diet assessment | Baseline, 1-month, 2-months, 5-months
  A bespoke measure developed for this project and the feasibility project, in consultation with people with coeliac disease and dietitians, to assess parent knowledge of the gluten-free diet. Scores range from 0-12, with higher scores indicating greater knowledge.
Gluten-free diet adherence (parent-report) | Baseline, 1-month, 2-months, 5-months
  Parent reported measure to assess children's gluten-free diet adherence, consisting of five levels (0-4). Levels 0 or 1 indicate poor diet adherence, 2 indicates moderate adherence, and 3-4 indicates strict adherence.
Gluten-free diet adherence (child-report, Biagi et al., 2009). | Baseline, 1-month, 2-months, 5-months
  Child reported measure to assess children's gluten-free diet adherence (optional) consisting of five levels (0-4). Levels 0 or 1 indicate poor diet adherence, 2 indicates moderate adherence, and 3-4 indicates strict adherence.
Warwick-Edinburgh Mental Wellbeing scale | Baseline, 1-month, 2-months, 5-months
  The scale has 14 items assessing various aspects of mental wellbeing. Scores range from 14 to 70, reflecting greater mental wellbeing with higher scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Surrey County Hospital, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wood JJ, McLeod BD, Sigman M, Hwang WC, Chu BC. Parenting and childhood anxiety: theory, empirical findings, and future directions. J Child Psychol Psychiatry. 2003 Jan;44(1):134-51. doi: 10.1111/1469-7610.00106. PMID 12553416
- [Background] White LE, Bannerman E, Gillett PM. Coeliac disease and the gluten-free diet: a review of the burdens; factors associated with adherence and impact on health-related quality of life, with specific focus on adolescence. J Hum Nutr Diet. 2016 Oct;29(5):593-606. doi: 10.1111/jhn.12375. Epub 2016 May 23. PMID 27214084
- [Background] Majewska Z, Dilling-Ostrowska E. [Speech disorders in childhood]. Psychiatr Neurol Med Psychol Beih. 1970;13-14:94-9. German. PMID 4143528
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Silvester JA, Weiten D, Graff LA, Walker JR, Duerksen DR. Living gluten-free: adherence, knowledge, lifestyle adaptations and feelings towards a gluten-free diet. J Hum Nutr Diet. 2016 Jun;29(3):374-82. doi: 10.1111/jhn.12316. Epub 2015 Apr 20. PMID 25891988
- [Background] Satherley RM, Coburn SS, Germone M. The Impact of Celiac Disease on Caregivers' Well-being: An Integrative Review. J Pediatr Gastroenterol Nutr. 2020 Mar;70(3):295-303. doi: 10.1097/MPG.0000000000002572. PMID 31789773
- [Background] Russo C, Wolf RL, Leichter HJ, Lee AR, Reilly NR, Zybert P, Green PHR, Lebwohl B. Impact of a Child's Celiac Disease Diagnosis and Management on the Family. Dig Dis Sci. 2020 Oct;65(10):2959-2969. doi: 10.1007/s10620-020-06316-0. Epub 2020 May 15. PMID 32415563
- [Background] Guedes NG, Silva LAD, Bessa CC, Santos JCD, Silva VMD, Lopes MVO. Anxiety and depression: a study of psychoaffective, family-related, and daily-life factors in celiac individuals. Rev Bras Enferm. 2020 Sep 21;73Suppl 1(Suppl 1):e20200086. doi: 10.1590/0034-7167-2020-0086. eCollection 2020. English, Portuguese. PMID 32965317
- [Background] Jones CJ, Read R, O'Donnell N, Wakelin K, John M, Skene SS, Stewart R, Hale L, Cooke D, Kanumakala S, Satherley RM. PRIORITY Trial: Results from a feasibility randomised controlled trial of a psychoeducational intervention for parents to prevent disordered eating in children and young people with type 1 diabetes. Diabet Med. 2024 Apr;41(4):e15263. doi: 10.1111/dme.15263. Epub 2023 Dec 15. PMID 38100228
- [Background] Jones CJ, O'Donnell N, John M, Cooke D, Stewart R, Hale L, Skene SS, Kanumakala S, Harrington M, Satherley RM. PaRent InterventiOn to pRevent dIsordered eating in children with TYpe 1 diabetes (PRIORITY): Study protocol for a feasibility randomised controlled trial. Diabet Med. 2022 Apr;39(4):e14738. doi: 10.1111/dme.14738. Epub 2021 Nov 12. PMID 34741779
- [Background] Jordan NE, Li Y, Magrini D, Simpson S, Reilly NR, Defelice AR, Sockolow R, Green PH. Development and validation of a celiac disease quality of life instrument for North American children. J Pediatr Gastroenterol Nutr. 2013 Oct;57(4):477-86. doi: 10.1097/MPG.0b013e31829b68a1. PMID 23689265
- [Background] Mazzone L, Reale L, Spina M, Guarnera M, Lionetti E, Martorana S, Mazzone D. Compliant gluten-free children with celiac disease: an evaluation of psychological distress. BMC Pediatr. 2011 May 27;11:46. doi: 10.1186/1471-2431-11-46. PMID 21619651
- [Background] Olsson C, Lyon P, Hornell A, Ivarsson A, Sydner YM. Food that makes you different: the stigma experienced by adolescents with celiac disease. Qual Health Res. 2009 Jul;19(7):976-84. doi: 10.1177/1049732309338722. PMID 19556403
- [Background] Biagi F, Andrealli A, Bianchi PI, Marchese A, Klersy C, Corazza GR. A gluten-free diet score to evaluate dietary compliance in patients with coeliac disease. Br J Nutr. 2009 Sep;102(6):882-7. doi: 10.1017/S0007114509301579. Epub 2009 Mar 31. PMID 19331704